CLINICAL TRIAL: NCT01286909
Title: Trial of Laflavon in Patients With Metabolic Syndrome to Evaluate Its Effectiveness in Lowering Triglycerides and Raising High-Density Lipoprotein (HDL)
Brief Title: Efficacy of Laflavon in Lowering Triglycerides and Raising High-Density Lipoprotein (HDL)
Acronym: LaFlavon
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omicron Pharmaceuticals (Industry)
Responsible Party: Dr. Akram Echtay, Omicron Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP912011
Record Dates: First submitted 2011-01-09; First posted 2011-01-31 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Metabolic Disease
Keywords: Metabolic
MeSH Terms: conditions — Metabolic Diseases | interventions — Lycopene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LaFlavon (Experimental)
  Interventions: Dietary Supplement: LaFlavon
- Placebo (No Intervention)

INTERVENTIONS:
Dietary Supplement: LaFlavon — two tablets of LaFlavon (two x 3.5mg lycopene/25 mg soy isoflavone) daily for three months
  Other Names: Lycopene/Isoflavon
  Arms: LaFlavon

SUMMARY:
A trial of LaFlavon in Patients with Metabolic Syndrome to Evaluate its Effectiveness in Lowering Triglycerides and Raising High-Density Lipoprotein (HDL).

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women with Metabolic Syndrome
2. Elevated Triglycerides (> 150)
3. Low High-Density Lipoprotein (HDL) (< 35)
4. Willingness to take study nutritional supplement once a day for 3 months

Exclusion Criteria:

1. Women who are pregnant, nursing, or who intend pregnancy during the period of treatment
2. Known milk, soy or whey allergy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Increase in High-Density Lipoprotein (HDL) | Change from Baseline in High-Density Lipoprotein (HDL) at 3 months

SECONDARY OUTCOMES:
changes of liver enzymes | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Akram Echtay, M.D., Principal Investigator — Rafic Hariri University Hospital
Locations (1):
- Rafic Hariri University Hospital, Beirut, Lebanon